CLINICAL TRIAL: NCT02230228
Title: A Phase 1, Open Label, Repeat Dose Study to Investigate the Safety and Pharmacokinetics of 4-week Daily Dosing of ALK-001 in Healthy Volunteers
Brief Title: Phase 1 Safety Study of ALK-001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkeus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALK001-P1001
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Stargardt Disease; Age-related Macular Degeneration; Other Retinal Dystrophies
MeSH Terms: conditions — Stargardt Disease; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALK-001 capsules (Experimental)
  Interventions: Drug: ALK-001 (No generic name)

INTERVENTIONS:
Drug: ALK-001 (No generic name) — Daily, oral administration of ALK-001 capsules.
  Other Names: C20-D3-Retinyl Acetate; C20 Deuterated vitamin A

SUMMARY:
This protocol is a phase 1 clinical study to assess the safety and pharmacokinetics of ALK-001 in healthy volunteers. Please contact trials@alkeus.com for any questions.

ELIGIBILITY:
Main Inclusion Criteria

* Adult between 21 and 70 years old (inclusive)
* Healthy subject, as judged by investigator
* Subject is able and willing to comply with study requirements (study medication compliance, schedule of follow-up visits)
* Subject has provided informed consent to participate
* If female, subject uses a medically accepted birth control method and agrees to use such a method for entire clinical trial period

Main Exclusion Criteria:

* Subject has taken disallowed items during the past 30 days
* Female with a positive urine pregnancy test at screening
* Lactating woman
* Subject has participated in any clinical study involving an investigational drug, biologic or device, during the past 30 days
* History or current evidence of gastrointestinal malabsorption
* Subject has any other medical condition, which in the opinion of the investigator, is likely to prevent compliance with protocol and/or interfere with successful collection of study
* Subject has, in the opinion of investigator, clinically significant laboratory result(s), positive drug or alcohol screening, or ECG, which makes subject unsuitable for participation.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety of 4-week daily dosing of ALK-001 in healthy adults. | 4 weeks
  Safety evaluations combine: adverse events (AE), laboratory testing (hematology and biochemistry panels), 12-lead electrocardiograms (ECGs), vital signs, physical examination, and visual function (visual acuity and a self-reported questionnaire).